CLINICAL TRIAL: NCT03462836
Title: The Effects of Optimizing Post-operative Pain Management With Multi Modal Analgesia on Immune Suppression and Oncologic Outcome in Patients Undergoing Laparoscopic Colorectal Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The results of the primary endpoints of this study are expected to be difficult to identify, thus canceling the study to readjust the study plan.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4-2017-0773
Record Dates: First submitted 2018-02-06; First posted 2018-03-13 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Laparoscopic Colorectal Resection Due to Cancer
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IV ketamine/lidocaine/IV PCA (MA) group (Experimental): In addition to basic anesthetic methods, multimodal analgesia with IV ketamine, lidocaine and IV PCA apply
  Interventions: Drug: IV ketamine/lidocaine/IV PCA apply
- IV PCA only (CA) group (Active Comparator): In addition to basic anesthetic methods, only IC PCA apply for pain control
  Interventions: Drug: IV PCA only apply

INTERVENTIONS:
Drug: IV ketamine/lidocaine/IV PCA apply — In the MA group, 1.0 mg / kg of ketamine is diluted to a total volume of 10 ml. Slowly apply for 1 minute during surgical drape. 1 mg / kg of Lidocaine is loaded at the beginning of surgery. Lidocaine 1.5 mg / kg / hr is administered until the end of the operation.
  Arms: IV ketamine/lidocaine/IV PCA (MA) group
Drug: IV PCA only apply — IV PCA (fentanyl 10mcg/kg + nefopam (Acupan®) 80mg + Ramosetron (Nasea®) ) apply 30min before end of surgery.
  Arms: IV PCA only (CA) group

SUMMARY:
Traditionally, pain control methods based on narcotic analgesics have been used to control severe pain after surgery, but this has resulted in side effects such as vomiting, constipation, dizziness, mental confusion due to drugs, and respiratory depression. This slowed the recovery of the patient after surgery and increased the duration of hospitalization, which had a negative impact on the patient 's prognosis. In addition, research has been conducted on the use of various painkillers in a variety of ways over the past decade to reduce the dose of narcotic analgesics and to increase the effectiveness of pain control, since studies of anesthetics and narcotic analgesics have shown immunosuppressive effects.

This study investigate the effect of multimodal analgesics for postoperative pain control on immune function amd prognosis in patients undergoing laparoscopic colorectal cancer resection.

ELIGIBILITY:
Inclusion Criteria:

1. elective laparoscopic colorectal resection due to colorectal cancer
2. curative, resectable operation
3. ASA classification Ⅰ-Ⅲ

Exclusion Criteria:

1. elective co-operation due to distance metastasis
2. preoperative chemo/radiation therapy
3. drug allergy to opioid, tramadol, local anesthetics
4. MAOi medication (within 14 days of surgery)
5. decreased hepatic/renal function
6. Patients who can not read the consent form or are not fluent in Korean (illiterate, foreigner
7. pregnant, lactating women
8. palliative surgery

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2021-09-28 (Estimated)

PRIMARY OUTCOMES:
natural killer cell cytotoxicity | postoperative day #3
  Natural killer cell cytotoxicity is measured with NK Vue Kit™(ATGen, Gyeonggi-do, Korea).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, Republic of Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No